CLINICAL TRIAL: NCT03556475
Title: A Diagnostic Test to Develop an AECOPD Identification Tool Through Characteristic Variables Extracted From Diagnosed AECOPD Patients
Brief Title: Development of AECOPD Identification Tool (DETECT Study)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5252R00002
Record Dates: First submitted 2018-05-10; First posted 2018-06-14 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Acute Exacerbations of COPD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — This is an observational study and no samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Disease 1: Moderate to severe COPD Patients(n=90)
- Disease type 2-1): Patients with Mild/moderate AECOPD (n=60)
- Disease type 2-2): Patients with Severe AECOPD( n=60)
- Disease type 3: Non-COPD Patients with high risk factors (n=90)

SUMMARY:
This study is an observational, multi-center and cross sectional study,to develop an identification tool on purpose of differentiating COPD exacerbation from patients with respiratory symptoms in community hospitals of China.

DETAILED DESCRIPTION:
This is an observational, multi-center and cross-sectional study to develop an AECOPD identification tool. Estimated totally 7 tertiary hospitals with experts in respiratory area will be involved as the study sites. These study sites will cover the regions of China (Eastern, Southern, Northern, Central, Western and Northeastern region), to be representative for the patient features all over the country. The patients will be enrolled in a "consecutive" way, which is, the investigators will recruit the patients who are eligible and consented to participate in this study without personal tendency.

For the enrolled patients, a face to face visit between investigator and patient will be arranged. The evaluation for the symptoms and signs will be performed and the relevant data will be collected on the visit. In addition, other relevant tests (e.g. oxygen saturation, blood test, CAT, etc) and data (demographic, medical history, etc) will be collected on this visit.

ELIGIBILITY:
Inclusion Criteria:

-≥ 40 years old of age.

* Able to adequately understand written and verbal
* A signed and dated written informed consent must be obtained prior to the visits
* Patients see doctors due to suffering respiratory disease below:

Disease type 1 - diagnosed moderate and severe stable COPD

* Patients with a diagnosis of COPD and documented record with predicted ratio of FEV1 to forced vital capacity (FVC) < 0.70 before the study visit
* COPD with moderate to severe airflow obstruction (FEV1<0.8 predicted)

Disease type 2 - AECOPD

* Patients with a diagnosis of COPD and documented record with predicted ratio of FEV1 to forced vital capacity (FVC) < 0.70 before the study visit
* Patients consult the clinic or the emergency department because of acute worsening with an AECOPD (diagnosed by more than 2 clinical experts and refer to diagnosis criteria of Appendix 2)

Disease type 3

-Non-COPD patients with chronic respiratory symptoms such as cough, sputum and wheeze, dyspnea etc. (≥2 high risk factors )

Exclusion Criteria:

* Patients with severe cardiovascular disease, including uncontrolled hypertension with drug treatment, unstable angina, myocardial infarction within the last 6 months, NYHA class II congestive heart failure, severe arrhythmia, pericardial effusion, etc.
* Patients with lung cancer, esophageal cancer or mediastinal tumors;
* Patients who participated in any drug clinical trials within 4 weeks before enrollment;
* Patients with severe infection, indicated for intravenous antibiotics, antifungal or antiviral therapy;
* Patients suffering from mental illness and poor compliance;
* Patients inappropriate for inclusion decided by investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Disease type 1 : Moderate to severe COPD Patients(n=90); Disease type 2 : Patients with AECOPD
  a) Mild/moderate: n=60 c) Severe: n=60 Disease type 3 : Non-COPD Patients with high risk factors (n=90)
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Sensitivity(Sen) & Specificity(Spe) | Dec2017--Mar2020
  Each candidate factors will be tested and weighed. 6-8 factors are estimated to be identified and modelled to form AECOPD identification scale. The validity and efficacy of AECOPD identification tools will be assessed by internal verification.

CONTACTS AND LOCATIONS:
Overall Officials: Jian KANG, PhD, Principal Investigator — No 155. Nanjing street, Heping District, Liaoning Province
Locations (7):
- China (7):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Xi'an
  - Research Site, Xinxiang

REFERENCES:
- See also: CSR_Synopsis-DETECT.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5252R00002&attachmentIdentifier=99ec0663-fec8-4624-bf7e-4687d89e7726&fileName=CSR_Synopsis-DETECT.pdf&versionIdentifier=